CLINICAL TRIAL: NCT07140653
Title: Evaluation of Arcuate Incisions for Correcting Pre-Existing Corneal Astigmatism in Combination With the Light Adjustable Lens for Cataract and Refractive Lens Exchange Surgery
Brief Title: Arcuate Incisions With Light Adjustable Lens for Astigmatism Correction in Lens Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Center For Sight (Other)
Collaborators: LensAR Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFS 25-003
Record Dates: First submitted 2025-08-22; First posted 2025-08-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Femto arcs + LAL (Other)
  Interventions: Other: Femto arcs; Device: Light Adjustable Lens (LAL)

INTERVENTIONS:
Other: Femto arcs — Femtosecond laser-assisted arcuate corneal relaxing incisions (AK) will be performed to correct astigmatism.
Device: Light Adjustable Lens (LAL) — The LAL is intended to replace the natural lens at time of lens removal.

SUMMARY:
This study aims to evaluate the safety and effectiveness of femtosecond laser arcuate corneal relaxing incisions (AK) combined with Light Adjustable Lens (LAL) implantation for correcting pre-existing corneal astigmatism in patients undergoing cataract or refractive lens exchange surgery. Postoperative assessments will focus on residual refractive astigmatism, visual outcomes, patient satisfaction, and the incidence of adverse events. Arcuate keratotomy and toric IOLs are well-established methods for astigmatism correction, and this study will compare their combined effectiveness using advanced femtosecond laser technology.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be aged ≥ 21 years at the time of eligibility visit.
2. Subject must have a vector difference of 0.50 D or less in magnitude of pre-operative anterior corneal astigmatism as measured by the Pentacam AXL and the Zeiss IOLMaster 700 (Carl Zeiss Meditec).
3. Subject must be able and willing to comply with the study examination procedures.
4. Astigmatic treatment must require paired arcs <45mm in length.
5. Subject must be willing to complete the approved informed consent form.
6. Subject must have elected to undergo lens extraction and Light Adjustable Lens (LAL) implantation.
7. Subject must be willing and able to return for scheduled pre-op and follow-up examinations.
8. Subject must have central 7 mm of clear cornea without vascularization.

Exclusion Criteria:

1. Subject who has undergone previous corneal or intraocular surgery in the eye to be treated.
2. Subject with a history, signs or symptoms of ocular disease or atypical findings that would be contraindicated under standard of care for lens extraction surgery.
3. Subject with neuro-ophthalmic disease.
4. Diabetic or hypertensive subject with clinical evidence of retinal pathology that the investigator believes will significantly affect visual outcomes.
5. Subject with macular degenerative pathology identified at the preoperative visit that the investigator believes will significantly affect visual outcomes.
6. Subject with a history of steroid-responsive rise in intraocular pressure (IOP), preoperative IOP >25 mmHg, or uncontrolled glaucoma in either eye.
7. Subject with known lens/zonular instability.
8. Subject who cannot achieve dilated pupillary diameter > 6 mm.
9. Subject with abnormal corneal topography, including evidence of forme fruste keratoconus, keratoconus or pellucid marginal degeneration.
10. Subject with posterior segment disease or degeneration.
11. Subject with corneal disease or pathology that precludes an adequate view for imaging or transmission of laser wavelength of light.
12. Subject with known sensitivity to planned perioperative standard of care medications.
13. Subject participating in any other ophthalmic drug or device clinical trial during the time of this clinical assessment.
14. Subject with known sensitivity to planned assessment concomitant medications.
15. Subjects with severe dry eye syndrome (DES) or history of ocular inflammation that may impact visual outcomes.
16. Subject with irregular astigmatism in the eye to be treated.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of LAL adjustments required to achieve the desired refraction | 8 weeks after last lock-in

SECONDARY OUTCOMES:
Percentage of eyes with residual refractive astigmatism ≤ 0.50 D | 8 weeks after last lock-in

CONTACTS AND LOCATIONS:
Overall Officials: Priya Mathews, MD, Principal Investigator — Center For Sight - Clinical Studies
Locations (2):
- United States (2):
  - Center For Sight, Venice, Florida
  - Carolina Eyecare Physicians, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No